CLINICAL TRIAL: NCT00843817
Title: RhDNase Effect on Biodistribution of PMN Serine Proteases in Cystic Fibrosis Sputum
Brief Title: RhDNase and Biodistribution of PMN Serine Proteases in Cystic Fibrosis Sputum
Acronym: BioDNase
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PHAO08-PD BioDNase
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Last update posted 2022-03-16 (Actual); Status verified 2017-02

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — dornase alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DRUG (Experimental): PULMOZYME
  Interventions: Drug: Pulmozyme

INTERVENTIONS:
Drug: Pulmozyme — Pulmozyme® 2.5mg by inhalation

SUMMARY:
Serine proteases belonging to the elastase family are mainly responsible for lung tissue destruction as observed during cystic fibrosis. But anti-inflammatory therapies based on systemic or aerosolized protease-inhibitors administration, have not given the expected results until now. One reason would be the impaired access of therapeutic inhibitors to their molecular targets. It was recently shown that neutrophils actively secrete neutrophil extracellular traps (NETs) made of DNA that binds cationic proteases among other molecules. NETs together with DNA passively released from dead neutrophils contribute to the viscosity of CF expectorations which explains that rhDNase treatment fluidifies expectorations and improves the patient status. Preliminary experiments in our laboratory have shown that DNA degradation was associated with a significant increase of proteolytic activity in the sputum soluble fraction. However the efficacy of exogenous inhibitors is also improved in these conditions. Using the specific substrates and methodologies that we developed previously to measure cell-surface associated proteolytic activities, we will study the effects of DNase on the activity of individual proteases, their biodistribution in sputum and their regulation by potential therapeutic inhibitors. Enzymatic, immunochemical and microscopic (confocal and scanning) techniques will first be used for ex vivo studies on sputa freshly collected at the adult and paediatric CRCM in Tours, then on sputa from patients before and after administration of aerosolized rhDNase. We hypothesize that a better understanding of the biodistribution of neutrophil serine proteases and especially their binding to DNA will help designing new therapeutic strategies that facilitate inhibitor access to their protease targets.

ELIGIBILITY:
Inclusion Criteria:

* cystic fibrosis disease
* with rhDNase treatment

Exclusion Criteria:

* Acute push of the bronchopulmonary attack or hospitalization for treatment of the disease during 2 weeks previous
* Exposure to a antibiotherapy or treatment by corticoids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-04 (Actual); Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
The biodistribution of elastase, Protease 3 and cathepsine G in the expectorations will be measured by the management report of these proteases between the freezing fractionand the soluble fraction, before and after rhDNase administration. | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Patrice DIOT, PHD, Principal Investigator — University Hospital, Tours
Locations (1):
- University Hospital - Tours, Tours, France

IPD SHARING:
Plan to Share IPD: No